CLINICAL TRIAL: NCT04493632
Title: OncoSil Pancreatic Cancer Post-marketing Clinical REgistrY (OSPREY)
Brief Title: OSPREY is a Post-market, Global, Multicentre, Observational, Prospective Registry.
Acronym: OSPREY
Status: Recruiting | Type: Observational
Sponsor: OncoSil Medical Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: OSPREY01
Record Dates: First submitted 2020-07-21; First posted 2020-07-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Pancreatic Neoplasm; Digestive System Neoplasm; Neoplasms by Site; Neoplasms; Endocrine Gland Neoplasm; Digestive System Disease; Pancreatic Diseases; Endocrine System Diseases
Keywords: Pancreatic Cancer; Pancreas; Metastases; Pancreatic tumor; Unresectable; Locally advanced; Implantable; Radiographic; Device; Phosphorous-32; OncoSil™; Brachytherapy; Gemcitabine; Nab-paclitaxel; Abraxane
MeSH Terms: conditions — Pancreatic Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Endocrine Gland Neoplasms; Digestive System Diseases; Pancreatic Diseases; Endocrine System Diseases; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The OSPREY Patient Registry has been developed to collect and assess the performance and safety of the OncoSil™ device when used within the approved indication of unresectable, locally advanced pancreatic cancer, in combination with gemcitabine-based chemotherapy, within a real-world observational registry.

The Registry data will provide both complementary and contemporary information to the existing clinical data across various countries and will form part of the post-market clinical follow-up activities for OncoSil™. Therefore, the Registry will be implemented only in countries with regulatory (commercial) approval for the OncoSil™ device.

DETAILED DESCRIPTION:
OSPREY is a post-market, global, multicentre, observational, prospective registry in which data is recorded from patients who undergo OncoSil™ device implantation.

Countries intended for initial commercial distribution include Australia, Belgium, France, Germany, Italy, Singapore, Spain, & the United Kingdom.

Only patients who are intended to undergo treatment with the OncoSil™ device in the commercial (sales) setting will participate in this Registry.

Every patient who is prescribed OncoSil™ in the commercial setting will be approached by the Treating Physician to consent to participate in the OSPREY Patient Registry.

Patients who choose not to consent to participate in the OSPREY Patient Registry will not be excluded from being treated with the OncoSil™ device.

Five hundred patients (implanted with OncoSil™) will be recruited into the OSPREY Patient Registry. It is anticipated recruitment will be over a five-year period, subject to the rate of commercial adoption of the OncoSil™ device in the market.

To adequately collect data relating to the performance and safety of the OncoSil™ device, data will be collected from patients over a prescribed 12-month period from enrolment, the cohort is then followed to death or to 24-months post the date of the last enrolled patient implanted with OncoSil™.

Therefore, the Registry is expected to run for a seven-year period. Relevant observational data will be collected via medical record review.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed unresectable locally advanced pancreatic cancer (LAPC).
2. Patients who undergo OncoSil™ implantation at an eligible treatment facility.
3. Patients who have completed and signed the Patient Informed Consent Form (PICF) for the OSPREY Patient Registry.
4. Pancreatic target tumour recommended size of <7 cm (longest diameter) and <110 cc volume.
5. A clinically acceptable ECOG performance status.
6. Patients ≥ 18 years of age at screening.
7. To commence gemcitabine-based chemotherapy, (per Standard-of-Care are according to the approved prescribing schedule) post Registry enrolment.
8. Adequate biochemical tests, coagulation profile, haematological, renal, and hepatic function as determined by the Treating Physician.

Exclusion Criteria:

1. Patient Informed Consent Form (PICF) has not been completed and signed for the OSPREY Patient Registry.
2. Patients treated with OncoSil™ within an approved interventional clinical study (company or investigator-sponsored).
3. Evidence of distant metastases based on review of baseline CT scan.
4. More than one primary lesion.
5. In the opinion of the Treating Physician, EUS-directed implantation posing undue patient risk. This includes:

   * where previous EUS-FNA was considered technically too difficult to perform;
   * imaging demonstrates multiple collateral vessels surrounding or adjacent to the target tumour within the pancreas;
   * presence (or significant risk) of varices near to the target tumour.
6. Evidence of radiographic invasion into stomach or duodenum (if not certain, confirmation must be obtained prior to enrolment).
7. In the setting of recent, clinically significant pancreatitis, implantation is not recommended.
8. Pregnant or intending to commence a pregnancy within 12-months of the intended date of implantation or breastfeeding.
9. Patients who have a known history of hypersensitivity to silicon or phosphorous, or any of the OncoSil™ components

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patient who is intended to undergo implantation of the OncoSil™ device when used within the approved indication of unresectable, locally advanced pancreatic cancer, in combination with gemcitabine-based chemotherapy, in the commercial (sales) setting will be approached by the Treating Physician to consent to participate in the OSPREY Patient Registry.
  Patients who choose not to consent to participate in the OSPREY Patient Registry will not be excluded from being treated with the OncoSil™ device.
  .
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-04-12 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of Device | Followed to death or to 24-months post the date of the last enrolled patient implanted with OncoSil™
  The analysis for safety within the real-world setting will be performed. The safety of OncoSil™ is defined by the Adverse Event profile. All safety summaries will be produced for the Intention-To-Treat (ITT) population. Adverse events will be coded using Medical Dictionary for Regulatory Activities (MedDRA). All Adverse Events recorded during the Registry will be listed.
  Summary tables will be produced for Treatment Emergent Adverse Events (TEAEs). The number and percentage of patients with device-related Adverse Events by system organ class (SOC) and preferred term will be tabulated. Similar summaries will be produced by severity of event (both mild, moderate or severe, CTCAE grade 1-4) and drug and/or device relationship.
  In addition, summary tables will be produced for serious TEAEs and TEAEs associated with special interest acute/late radiation effects and or withdrawal.
Device Implantation Performance | 7 years
  Safety of the implantation of OncoSil™ within the target tumour will be measured by means of procedure-related Adverse Events. An assessment of the utility of OncoSil™ Implantation will be made and listed appropriately.
Overall Survival | Followed to death or to 24-months post the date of the last enrolled patient implanted with OncoSil™
  Overall survival (OS) is defined as the time from enrolment to the date of death from any cause. Patients who are alive or permanently lost to follow-up at the cut-off date for the analysis will be censored at the last date the patient was known to be alive.
  Overall Survival (OS) will be analysed at the interim analysis and once all 500 OncoSil™ implanted patients have been followed to death or to 24-months post the date of the last enrolled/treated patient.
tumour response as demonstrated by target tumour response demonstrated by RECIST 1.1 | 7 years
  Target (implanted) tumor response (local and distant)
Resection Rates | 7 years
  Surgical resection rates and outcome

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Ross, MRCP, MBBS, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust, London, UK
Locations (9):
- Spain (7):
  - Complejo Hospitalario Universitario Insular Materno-Infantil, Las Palmas de Gran Canaria
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario de Fuenlabrada, Madrid
  - Hospital Universitario Doce De Octobre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Clinica Universidad De Navarra, Pamplona
  - Hospital Clinico Universitario De Valladolid, Valladolid
- United Kingdom (2):
  - Hammersmith Hospital, London
  - The London Clinic, London

IPD SHARING:
Plan to Share IPD: No